CLINICAL TRIAL: NCT01774825
Title: Double-blind, Randomized, Placebo-controlled, Bicentric Clinical Investigation to Evaluate the Safety and Efficacy of IQP-CL-101 in the Symptomatic Improvement of Irritable Bowel Syndrome (IBS)
Brief Title: IQP-CL-101 in IBS Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INQ/028111
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — IQP-CL-101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IQP-CL-101 (Active Comparator): 2 softgels twice a day
  Interventions: Dietary Supplement: IQP-CL-101
- Placebo (Placebo Comparator): 2 softgels twice a day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-CL-101 — 2 softgels twice a day
  Arms: IQP-CL-101
Other: Placebo — 2 softgels twice a day
  Arms: Placebo

SUMMARY:
After 2 weeks of run-in period, subjects are randomized to either IQP-CL-101 or a matching placebo. Over 8 weeks, the subjects are monitored for improvements in IBS symptoms

ELIGIBILITY:
Inclusion Criteria:

* Fulfils Rome-III criteria for IBS diagnosis
* Females' agreement to use appropriate birth control methods during the active study period for females of childbearing potential
* Subject declares in writing his/her consent to participate, understands requirements of the study and is willing to comply

Exclusion Criteria:

* Known sensitivity to any of the ingredients of IQP-CL-101
* Clinically relevant abnormalities in colonoscopy within the last 2 years prior to randomization
* Other causes of IBS symptoms such as inflammatory bowel disease (IBD), microscopic colitis, celiac disease, history of abdominal obstruction, cholecystitis, pancreatitis, ileus, or any gastrointestinal bleeding
* Use of medications that could influence GI functions (e.g. antibiotics, laxatives, opioids, glucocorticoids, anticholinergics, or anti-diarrheals) within 1 month prior to randomization
* Clinically relevant excursions of safety parameters
* Any other conditions deemed relevant by the investigator(s)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
IBS-SSS (Severity Symptom Score) | 8 weeks
  The questionnaire is to be completed by the subject

SECONDARY OUTCOMES:
IBS-GIS (Global Improvement Score) | 8 weeks
  The questionnaire is to be completed by the subject
IBS-QOL (Quality of Life) | 8 weeks
  The questionnaire is to be completed by the subject
Pain and discomfort diary | 8 weeks
  The diary is to be completed by the subject on a daily basis
Efficacy assessment by investigator | 8 weeks
  The investigator rates the efficacy of the investigational product using a 4-point Likert scale (poor, moderate, good, very good)
Efficacy assessment by subject | 8 weeks
  The subject rates the efficacy of the investigational product using a 4-point Likert scale (poor, moderate, good, very good)
Full blood count | 8 weeks
  After sampling, venous blood samples will be transported on same day in cooler boxes to a central laboratory for analysis of hemoglobin, hematocrit, erythrocytes, thrombocytes, and leucocytes
Clinical chemistry | 8 weeks
  Venous blood samples are obtained at screening and the end of the study (8 weeks)
Fecal calprotectin | 8 weeks
  The samples will be later tested by an enzyme immunoassay (ELISA) specific for calprotectin
Blood pressure | 8 weeks
  Sitting blood pressure and heart rate will be measured using standard devices
Safety assessment by subject | 8 weeks
  The subject rates the safety of the IP using a 4-point Likert scale (poor, moderate, good, very good)
Safety assessment by investigator | 8 weeks
  The investigator rates the safety of the IP using a 4-point Likert scale (poor, moderate, good, very good)
Adverse events | 8 weeks
  At all visits, subjects will be asked if any AE has occurred; such events will be recorded in the source documents and case report forms

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grube, MD, Principal Investigator — Private Practice
Locations (1):
- Barbara Grube, Berlin, State of Berlin, Germany